CLINICAL TRIAL: NCT00911599
Title: A Prospective Randomized Clinical Trial Comparing Ion Levels and Clinical Outcomes of the CONSERVE® A-Class Total Hip System With BFH® Technology to Metal on Polyethylene Total Hip Replacement
Brief Title: RCT Comparing Ion Levels and Clinical Outcomes of A-Class BFH to Metal on Polyethylene Total Hip Replacement
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006-506
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Hip Joint; Osteoarthritis; Arthroplasty
Keywords: Individuals undergoing unilateral total hip replacement.
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conserve Total Hip with BFH (Active Comparator): CONSERVE® A-Class Total Hip with BFH technology. Blood and urine samples will be collected and blood metal ion levels will be analyzed and compared to samples from the other group.
  Interventions: Diagnostic Test: Blood metal ion levels
- Metal with Polyethylene Liner (Active Comparator): Metal on polyethylene total hip replacement. Blood and urine samples will be collected and blood metal ion levels will be analyzed and compared to samples from the other group.
  Interventions: Diagnostic Test: Blood metal ion levels

INTERVENTIONS:
Diagnostic Test: Blood metal ion levels — Blood and urine will be collected and the levels of cobalt and chromium ions will be tested.

SUMMARY:
The main purpose of this prospective randomized controlled trial is to compare the concentrations of metal ions in the blood and urine of patients receiving implants that are identical except for the acetabular component: one is a monoblock and all cobalt chrome, and the other is modular with a titanium acetabular shell with a polyethylene insert.

DETAILED DESCRIPTION:
The primary aim of this study is to demonstrate that blood ion levels (cobalt and chromium) are lower at one year in patients who receive a metal on polyethylene total hip as compared to CONSERVE® A-Class Total Hip with BFH® technology. Secondary aims include the gathering of clinical data regarding survival and dislocation rates at two years post surgery, as well as the assessment of pain, physical function, radiographic and clinical outcome at the two year interval.

ELIGIBILITY:
Inclusion Criteria:

* Individuals undergoing unilateral total hip replacement.
* Patients 50 to 70 years of age.

Exclusion Criteria:

* Patients who have previously undergone any type of joint replacement.
* Patients with evidence of active infection.
* Patients with a documented allergy to cobalt chromium molybdenum.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Metal ion levels | 24 months
  To compare the metal ion levels between the advanced metal system and the traditional metal on polyethylene total hip replacement system.

SECONDARY OUTCOMES:
Dislocation Rate | 24 months
  Radiographic images will be taken to evaluate dislocation rate
Complications | 24 months
  All complications will be continually recorded.
Change in Harris Hip Score | 24 months
  Hip disability will be assessed using the Harris Hip Score. The questionnaire is one of the most commonly used hip scores for assessment of hip function. It comprises of 10 sections: Pain, Support, Limp, Distance walked, Stairs, Public Transportation, Sitting, Putting on Shoes/Socks, Presence of Deformity and Range of Motion (flexion, extension, abduction, adduction, internal and external rotation. The score of these items are summed together to get the total score. Scoring can range from 0 to 100. Scores less then 70 are poor, scores 70 to 79 are fair, scores 80 to 89 are good, and scores 90 to 100 are excellent.
Change in RAND-36 Health Survey | 24 months
  Health status will be assessed using the RAND-36 Health Survey. The survey contains eight concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item referring to a perceived change in health. A high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range. The lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved.
Change in UCLA Questionnaire | 24 months
  Patient-reported activity level will be assessed using the UCLA questionnaire. The index is self-administered and assesses current activity level. The UCLA scale is a simple scale ranging from 1 to 10. A low number (1) signifies very low activity levels, whereas 10 signifies a high activity level. One number is selected to best reflect the participants current activity level.
Change in WOMAC Questionnaire | 24 months
  Patient-reported hip functionality will be assessed using the WOMAC questionnaire. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is widely used as a standard assessment of arthritis in the hip joint. The Index is self-administered and assesses the three dimensions of pain (5 items), joint stiffness (2 items), and Physical Function (17 items) in hip osteoarthritis using 24 questions. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme. These correspond to an ordinal scale of 0-4. Scores are summed with higher scores indicating worse pain, stiffness, and function.

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Beaule, MD, FRCSC, Principal Investigator — University of Ottawa / The Ottawa Hospital
Locations (1):
- Ottawa Hospital - General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gofton W, Beaule PE. Serum Metal Ions with a Titanium Modular Neck Total Hip Replacement System. J Arthroplasty. 2015 Oct;30(10):1781-6. doi: 10.1016/j.arth.2015.04.040. Epub 2015 May 9. PMID 26027522
- [Result] Beaule PE, Kim PR, Hamdi A, Fazekas A. A prospective metal ion study of large-head metal-on-metal bearing: a matched-pair analysis of hip resurfacing versus total hip replacement. Orthop Clin North Am. 2011 Apr;42(2):251-7, ix. doi: 10.1016/j.ocl.2011.01.005. PMID 21435499